CLINICAL TRIAL: NCT06010875
Title: A Phase I Clinical Study to Assess the Safety and Efficacy of CD70-targeted CAR-T in the Treatment of CD70-positive Advanced/Metastatic Solid Tumors
Brief Title: A Clinical Research About CD70-targeted CAR-T in the Treatment of CD70-positive Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Collaborators: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBC052
Record Dates: First submitted 2023-08-18; First posted 2023-08-25 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-08

CONDITIONS: Renal Cell Carcinoma; Ovarian Cancer; Cervix Cancer; Metastatic Cancer; Advanced Cancer
Keywords: CAR-T; CD70
MeSH Terms: conditions — Carcinoma, Renal Cell; Ovarian Neoplasms; Uterine Cervical Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous of CD70-targeted CAR-T (Experimental): Infusion of CD70-targeted CAR-T cells by dose of 1-10x10^6 cells/kg
  Interventions: Biological: CD70 CAR-T cells
- intraperitoneal injection of CD70-targeted CAR-T (Experimental): Infusion of CD70-targeted CAR-T cells by dose of 1-10x10^6 cells/kg
  Interventions: Biological: CD70 CAR-T cells

INTERVENTIONS:
Biological: CD70 CAR-T cells — After lymphodepletion with Fludarabine and Cyclophosphamide,CAR T cells were transfused intravenically
  Arms: Intravenous of CD70-targeted CAR-T
Biological: CD70 CAR-T cells — After lymphodepletion with Fludarabine and Cyclophosphamide,CAR T cells were injected intraperitoneally
  Arms: intraperitoneal injection of CD70-targeted CAR-T

SUMMARY:
This is a single-center, double-arm, open-label study. this study plans to evaluate the safety and efficacy of CD70-targeting CAR-T cells in the treatment of CD70-positive advanced/metastatic solid tumors, and obtain recommended doses and infusion patterns.

DETAILED DESCRIPTION:
The research designs to follow 2 groups：Intravenous infusion group and Intraperitoneal injection group；each group sets up 2 phases,the first phase is dose discovery phase to obtain recommended doses,the second phase is dose expansion phase to verify the safety in the recommended doses. In the discovery phase,each group puts up 4 dose groups, adopting a dose-escalating 3+3 design, and plan to recruit about 12 subjects with CD70-positive advanced/metastatic solid tumors.In the dose expansion phase,each group will choose one or two dose groups to verify the safety and efficacy at this dose,and plan to recruit about 6 subjects in each dose group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female;
2. Advanced/metastatic solid tumor confirmed by histopathology or cytology (paraffin section or fresh biopsy tumor tissue specimen) (positive tumor CD70 expression (tumor CD70 positive (IHC 3+) confirmed by histology or pathology)) ;
3. At least after TKI/PARPi, anti-vascular drug treatment is ineffective, there is no available standard treatment plan or standard treatment fails or intolerable (disease progression or intolerance such as surgery, chemotherapy, radiotherapy, targeted therapy, etc.), There is currently no effective treatment;
4. Measurable and evaluable lesions defined by RECIST version 1.1: Measurable disease is defined as at least one lesion that can be accurately measured on at least one level (long diameter needs to be recorded); ), when measured by magnetic resonance imaging (MRI), each lesion must be >10mm, The lymph node must be >15mm in the short axis;
5. ECOG 0-2 points (Appendix 2);
6. The expected survival time is more than 12 weeks;
7. No serious mental disorder;
8. The functions of important organs are basically normal:

   1. Hematopoietic function: neutrophils 1.0×109/L, platelets 75×109/L, hemoglobin 80g/L;
   2. Cardiac function: echocardiography showed cardiac ejection fraction ≥50%, and no obvious abnormality was found on electrocardiogram;
   3. Renal function: serum creatinine≤2.0×ULN;
   4. Liver function: ALT and AST ≤2.0×ULN (for patients with liver tumor infiltration, it can be relaxed to ≤3.0×ULN);
   5. Total bilirubin ≤2.0×ULN (Gilbert syndrome or combined liver tumor infiltration can be relaxed to ≤3.0×ULN);
   6. Oxygen saturation > 92% in non-oxygen state.
9. Have apheresis or venous blood collection standards, and have no other contraindications for cell collection;
10. Subjects agree to use reliable and effective contraceptive methods for contraception within 1 year after signing the informed consent form to receiving CAR-T cell infusion (excluding rhythm contraception);
11. Subjects or their guardians agree to participate in this clinical trial and sign the ICF, indicating that they understand the purpose and procedures of this clinical trial and are willing to participate in the research.

Exclusion Criteria:

1. Received anti-CD70 drug treatment before screening;
2. Active/symptomatic central nervous system metastases or meningeal metastases at the time of screening; subjects with brain metastases who have been treated must be confirmed to have no imaging evidence of progression ≥ 4 weeks after the end of treatment before they can be enrolled;
3. Received any of the following treatments before screening:

   1. Participated in other interventional clinical studies before screening, including: the last use of unmarketed new drugs is less than 3 months before cell reinfusion, or the last use of marketed drugs is less than 5 half-lives from cell reinfusion;
   2. Received anti-tumor therapy such as chemotherapy and targeted therapy within 2 weeks or at least 5 half-lives (whichever is shorter) before apheresis;
   3. Received systemic corticosteroid therapy at doses greater than 10 mg/day prednisone (or equivalent doses of other corticosteroids) within 2 weeks prior to apheresis (inhalation or topical allowed in the absence of active autoimmune disease Use steroids and adrenal corticosteroid replacement at doses greater than 10 mg/day of prednisone);
   4. Received live attenuated vaccine within 4 weeks before screening;
4. Active infection or uncontrollable infection requiring systemic treatment within 1 week before screening;
5. Malignant tumors other than the target tumor within 3 years before screening, except for the following: malignant tumors that have received radical treatment, and no known active disease within ≥ 3 years before enrollment; or Treated non-melanoma skin cancer with no evidence of disease;
6. Suffering from any of the following heart diseases:

   1. New York Heart Association (NYHA) stage III or IV congestive heart failure;
   2. Myocardial infarction or coronary artery bypass grafting (CABG) within 6 months before enrollment;
   3. Clinically significant ventricular arrhythmia, or a history of unexplained syncope (except those caused by vasovagal or dehydration);
   4. History of severe nonischemic cardiomyopathy.
7. Known to have active or uncontrolled autoimmune diseases, such as Crohns disease, rheumatoid arthritis, systemic lupus erythematosus, systemic vasculitis, etc.;
8. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer detection is greater than the normal range; hepatitis C virus (HCV) antibody positive and peripheral blood type C Hepatitis virus (HCV) RNA titer detection greater than normal range Human immunodeficiency virus (HIV) antibody positive; syphilis positive test; cytomegalovirus (CMV) DNA test positive;
9. The subject has experienced venous thromboembolic events (for example: pulmonary embolism) and still needs anticoagulation therapy, or meets the following conditions: a. Bleeding with grades 3 to 4 for more than 30 days; b. There are venous Sequelae caused by embolism (such as persistent dyspnea and hypoxia); Arterial embolism but those who do not meet the above conditions can participate in the trial);
10. Poorly controlled hypertension, defined as systolic blood pressure ≥150mmHg and/or diastolic blood pressure ≥90mmHg (blood pressure values are measured based on the average of 3 readings at least 2 minutes apart, blood pressure ≥150/90mmHg at initial screening Receive antihypertensive treatment, if the treatment is well controlled and blood pressure is less than 150/90mmHg, screening can be performed);
11. Women who are pregnant or breastfeeding, and male or female subjects who plan to have children within 1 year after receiving CAR-T cell reinfusion;
12. Other investigators deem it unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events after CD70 CAR-T cells infusion [Safety and Tolerability] | 28 days
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
Obtain the maximum tolerated dose of CD70 CAR-T cells[Safety and Tolerability] | 28 days
  Dose-limiting toxicity after cell infusion

SECONDARY OUTCOMES:
Disease control rate of CAR-T cell preparations in CD70 positive advanced malignancies [Effectiveness] | 3 months
  Disease control rate: The proportion of subjects who achieved CR, PR, SD after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Objective response rate (ORR) of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 3 months
  Objective response rate includes：The proportion of subjects who achieved CR, PR after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Duration of Response (DOR) of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 2 years
  DOR will be assessed from the first assessment of CR/PR/SD to the first assessment of recurrence or progression of the disease or death from any cause
Progress-free survival(PFS) of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 2 years
  PFS will be assessed from the first CD70-CAR-T cell infusion to death from any cause or the first assessment of progression(Assessed based on RECIST criteria)
Overall survival(OS)of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 2 years
  OS will be assessed from the first CD70-CAR-T cell infusion to death from any cause (Assessed based on RECIST criteria)
AUCS of CD70 CAR-T cells [Cell dynamics] | 3 months
  AUCS is defined as the area under the curve in 90 days
CMAX of CD70 CAR-T cells [Cell dynamics] | 3 months
  CMAX is defined as the highest concentration of CD70 CAR-T cells expanded in peripheral blood
TMAX of CD70 CAR-T cells[Cell dynamics] | 3 months
  TMAX is defined as the time to reach the highest concentration
Pharmacodynamics of CD70 CAR-T cells[Cell dynamics] | 3 months
  Concentration levels of CAR-T-related serum cytokines such as CRP, IL-6, ferritin at each time point，which measured by Chemiluminescence method

OTHER OUTCOMES:
The correlation between CD70 positive rate and safety | 2 years
  assessment the correlation between CD70 positive rate and the incidence of CRA and ICANS
Correlation between CD70 positive rate and efficacy | 2 years
  assessment the correlation between CD70 positive rate and the disease control rate，Disease control rate: including CR, PR and SD
Overall survival(OS)of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 2 years
  OS will be assessed from the first CD70-CAR-T cell infusion to death from any cause (Assessed by investigators based on IRECIST criteria)
Progress-free survival(PFS) of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 2 years
  PFS will be assessed from the first CD70-CAR-T cell infusion to death from any cause or the first assessment of progression (Assessed by investigators based on IRECIST criteria)
Duration of Response (DOR) of CD70 CAR-T treatment in patients with CD70-positive advanced malignancies[Effectiveness] | 2 years
  DOR will be assessed from the first assessment of CR/PR/SD to the first assessment of recurrence or progression of the disease or death from any cause (Assessed by investigators based on IRECIST criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, M.D, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China